CLINICAL TRIAL: NCT03474211
Title: Prevalence of HPV Infection Using Self-sampling Screening and Monitoring the Earlier Impact of HPV-Vaccination Program in Switzerland
Brief Title: Prevalence of HPV Infection Using Self-sampling
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jeannot Emilien, Principal Investigator, University Hospital, Geneva
Other Study IDs: CER: 15-257
Record Dates: First submitted 2018-02-21; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: HPV - Anogenital Human Papilloma Virus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vaccinated
- non vaccinated

SUMMARY:
Background: Currently prevalence of HPV infections for high risk strains among young women in Switzerland is unknown. In addition, since 2008 a vaccination program to prevent these infections has been implemented in a number of cantons, but its actual population impact is currently unknown. For now, HPV screening in Switzerland is mainly performed by gynecologists or during gynecological consultation at hospital. This method is certainly effective, but expensive; population coverage of screening is still insufficient. A whole segment of the target population does not participate in this screening especially young people of foreign origin, for various reasons: economic cost, no gynecological, and for other reasons.

Several studies raise the effectiveness and efficiency of self-sampling to increase coverage of screening, and the rate of participation of non-participants. Through this study, the investigators evaluate effectiveness of this vaccination on the prevalence of HPV infections using HPV prevalence kit and assess evolution of infection and clearance of HPV virus during 5 years in a population of young unvaccinated and vaccinated women.

Method: During the study, each participants will perform a vaginal swab sampling by auto to research HPV. These samples will be sent to a laboratory where HPV typing is done by PCR using the Anyplex ™ II technology.

The study will focus on a sample of 400 young women. Participants must complete a questionnaire containing demographic questions and their HPV immunization status. Vaccination coverage expected in this population is about 50%. Depending on the state of vaccination, two different groups will be vaccinated vs unvaccinated (200 women per group). The cases of HPV infection are then calculated for each group and compared as a function of the status of vaccination. Statistical tests will be applied McNemar's test for comparison between the HPV prevalence rates between the 2 groups.

Expected Results: This study will allow us to confirm the possibility of using self-sampling as a method of screening and monitoring of HPV infections in the general population, it will also enable us to document the effectiveness of HPV vaccination by comparing prevalence rate of HPV infections among a group of young girls vaccinated and not vaccine and assess evolution of infection and clearance of HPV virus.

ELIGIBILITY:
Inclusion Criteria:

* • Eligible women aged between 18-31 years attending of Haute Ecole de Santé - Genève and Faculty of Medicine at the University of Geneva.

  * Understands study procedures and accepts voluntarily to participate by signing the informed consent form (ICF)

Exclusion Criteria:

* • History of hysterectomy or treatment on the cervix during the last 12 months

Ages: 18 Years to 31 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: It will take place in the health school of health and Faculty of Medicine at the University of Geneva. Trial information on the University website will be available; it will also contain a phone number for helpline. Cards to check eligibility, registration and scheduling will be available. The HPV self-collection kit will be directly distributed to participants at the end of their courses to School of Health and University of Geneva School of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
To determine the HPV prevalence of vaccine-type: 19 high-risk HPV types and 9 low-risk HPV types in a population of young unvaccinated and vaccinated women | 1.5 years
  Number of unvaccinated and vaccinated women infected by an HPV virus as assessed by using self sampling HPV kit.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amadane M, de Pree C, Viviano M, Vassilakos P, Jeannot E, Petignat P. Characteristics of HPV-unvaccinated undergraduate health students in Switzerland, a cross sectional study. Arch Public Health. 2019 Jun 18;77:29. doi: 10.1186/s13690-019-0348-y. eCollection 2019. PMID 31236272

DOCUMENTS (1):
  • Study Protocol (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT03474211/Prot_000.pdf